CLINICAL TRIAL: NCT06575127
Title: Modified FOLFOXIRI Plus Target Therapy as a First Line Treatment for Advanced Colorectal Cancer a Prospective Phase Two Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdelaziz, Specialist of Oncology, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FOXIRI
Record Dates: First submitted 2024-08-25; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Neoplasm Malignant; Colon Cancer Stage 4
Keywords: Colon Cancer; MCRC; FOLFOXIRI
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms | interventions — FOLFOXIRI protocol; Panitumumab; Bevacizumab; Cetuximab

STUDY DESIGN:
Intervention Model Description: Phase II single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- modified FOLFOXIRI plus target therapy (Experimental): * Pre-Treatment Medications:
    1. Atropine SC: Administered before irinotecan infusion to prevent side effects.
    2. High-Risk Anti-Emetics Regimen: Used to prevent acute and delayed vomiting.
  * Chemotherapy Regimen: All eligible patients will receive the modified FOLFOXIRI regimen as follows:
    * Oxaliplatin: 85 mg/m² IV over 2 hours (Day 1)
    * Irinotecan: 150 mg/m² IV over 90 minutes (Day 1)
    * 5-FU: 2400 mg/m² IV over 48 hours infusion (Days 1)
  * Targeted Therapy: Administered according to NRAS/KRAS status and the location of the primary tumor:
    * KRAS/NRAS/BRAF Wild-Type (Left-Sided Tumor): Anti-EGFR treatment with either Panitumumab (6 mg/kg over 60 minutes, Day 1) or Cetuximab (500 mg/m², Day 1).
    * KRAS/NRAS Mutant or Right-Sided Tumor: Bevacizumab at a dose of 5 mg/kg IV over 30 to 90 minutes (Day 1).
  * Treatment Schedule: The treatment will be administered biweekly for a maximum of 12 cycles (6 months).
  Interventions: Drug: FOLFOXIRI Protocol

INTERVENTIONS:
Drug: FOLFOXIRI Protocol — as mentioned in Arm description
  Other Names: Panitumumab; Bevacizumab; Cetuximab; modified FOLFOXIRI

SUMMARY:
This prospective Phase II study aims to evaluate the efficacy and safety of a modified FOLFOXIRI regimen in the treatment of metastatic colorectal cancer (MCRC). FOLFOXIRI, though effective, is known for its high toxicity, necessitating close monitoring and dose adjustments. .

The primary endpoint is to assess the impact on the objective response rate and evaluate both acute and delayed toxicity. The secondary endpoints include studying the treatment's effectiveness as conversion therapy, along with disease-free survival (DFS) and overall survival (OS). The tertiary endpoint focuses on evaluating predictive and prognostic factors of significance.

This study seeks to balance the efficacy of FOLFOXIRI with a modified dose to minimize toxicity while maintaining therapeutic benefits, providing a potentially safer and effective option for patients with MCRC.

DETAILED DESCRIPTION:
This prospective Phase II clinical trial aims to assess the efficacy and safety of a modified dose regimen of FOLFOXIRI in the treatment of metastatic colorectal cancer (MCRC). FOLFOXIRI is a chemotherapy regimen known for its high toxicity, necessitating close monitoring, dose reductions, and supportive treatments. While previous studies have demonstrated the clinical efficacy of FOLFOXIRI compared to FOLIRI or FOLFOX, the regimen's toxicity remains a significant concern.

Intervention:

Modified FOLFOXIRI Regimen:

Oxaliplatin: 85 mg/m² IV over 2 hours (Day 1) Irinotecan: 150 mg/m² IV over 90 minutes (Day 1) 5-FU: 2400 mg/m² IV over 48 hours infusion (Day 1)

Targeted Therapy:

KRAS/NRAS/BRAF Wild-Type (Left-Sided Tumor): Anti-EGFR treatment with either Panitumumab (6 mg/kg IV over 60 minutes, Day 1) or Cetuximab (500 mg/m² IV, Day 1).

KRAS/NRAS Mutant or Right-Sided Tumor: Bevacizumab (5 mg/kg IV over 30-90 minutes, Day 1).

Treatment Schedule: Administered biweekly for a maximum of 12 cycles (6 months).

G-CSF Prophylaxis: Administered as primary prophylaxis for patients older than 55 and as secondary prophylaxis for those who develop grade ≥3 neutropenia.

Dose Modifications and Treatment-Related Toxicity:

Toxicity will be evaluated after each cycle using the Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0 (National Cancer Institute, 2017).

Dose Reduction Guidelines: A 25% dose reduction will be implemented for specific grade III/IV acute toxicities including neutropenia, febrile neutropenia, thrombocytopenia, diarrhea, mucositis/stomatitis, hand-foot syndrome, peripheral neuropathy, elevated liver enzymes, severe fatigue, hypertension, proteinuria, and dermatologic toxicity.

Treatment Discontinuation: Patients who experience further grade III/IV acute toxicity after dose reduction will be excluded from the study.

Treatment Duration:

Eligible for Surgery: Patients with a favorable response will receive a maximum of 8 cycles before surgical evaluation.

Ineligible for Surgery: Treatment will continue until the completion of 12 cycles, intolerable toxicity, or a maximum duration of 6 months.

Assessments:

Disease Assessment: Performed every 4 cycles (8 weeks) during the induction phase, followed by every 3 months. Quality of life will be evaluated using the EORTC QLQ C30 and CR 29 questionnaires.

Response Assessment: Based on RECIST v1.1 criteria, categorized as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD).

Statistical Analysis:

Survival Analysis: Kaplan-Meier estimates with one-sided log-rank tests will be used to analyze progression-free survival (PFS). Overall survival (OS) will be calculated from the date of histological diagnosis to the date of last follow-up or death.

Data Analysis: Data will be analyzed using IBM SPSS version 26. Quantitative data will be presented as means, standard deviations, and ranges, or as medians with interquartile ranges, depending on distribution. Qualitative data will be presented as frequencies and percentages. Chi-square tests will compare groups with qualitative data. The confidence interval is set at 95%, with a significance threshold of p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed unrespectable or metastatic colorectal cancer with or without primary tumor in situ.

* Patients were required to have measurable disease according to RECIST v1.1 (Response Evaluation Criteria in Solid Tumors) (Eisenhauer EA,2009)
* ECOG PS 0-1 better to exclude PS II as this protocol is known to be toxic
* Adequate baseline hematology and clinical chemistry labs
* Adequate cardiac function

Exclusion Criteria:

* Double Malignancy
* DPYD mutant patients
* Peripheral neuropathy grade 3 or higher patient due to other comorbidities
* Inflammatory bowel syndrome or any other chronic GIT disease
* Prior exposure to chemotherapy treatment for colorectal cancer in the metastatic setting
* Patients who have contraindications for one or more of the study protocol drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Treatment-related adverse events | 12 months
  evaluate treatment-related acute and delayed toxicity
Objective Response Rate | 6 months
  To assess the impact of the treatment on the objective response rate

SECONDARY OUTCOMES:
Conversion therapy | 4 months
  To assess the treatment's efficacy as a conversion therapy, transforming initially unresectable tumors to resectable ones, response rates will be evaluated every 4 treatment cycles according to RECIST v1.1 (Eisenhauer EA, 2009):
  Complete Response (CR): Disappearance of all lesions and pathological lymph nodes.
  Partial Response (PR): ≥30% decrease in the sum of the longest diameters (SLD) of target lesions, no new lesions, and no progression in non-target lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  Progressive Disease (PD): ≥20% increase in SLD or the appearance of new lesions.
  Patients eligible for surgery may receive up to 8 cycles before surgical evaluation. Those showing favorable response will be referred for potential surgical intervention.
Progression free survival | 12 months
  to study the impact of treatment on progression free survival
Overall survival | 24 months
  to study the impact of treatment on overall survival

OTHER OUTCOMES:
Prognostic and predictive values | 24 month
  To evaluate predictive and prognostic factors of significance and its impact ORR, PFS and OS

CONTACTS AND LOCATIONS:
Locations (1):
- Al Hussien University Hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
study protocol and statistical analysis will be shared

REFERENCES:
- [Background] Kalyan A, Kircher S, Shah H, Mulcahy M, Benson A. Updates on immunotherapy for colorectal cancer. J Gastrointest Oncol. 2018 Feb;9(1):160-169. doi: 10.21037/jgo.2018.01.17. PMID 29564182
- [Result] Amado RG, Wolf M, Peeters M, Van Cutsem E, Siena S, Freeman DJ, Juan T, Sikorski R, Suggs S, Radinsky R, Patterson SD, Chang DD. Wild-type KRAS is required for panitumumab efficacy in patients with metastatic colorectal cancer. J Clin Oncol. 2008 Apr 1;26(10):1626-34. doi: 10.1200/JCO.2007.14.7116. Epub 2008 Mar 3. PMID 18316791
- [Result] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Result] Douillard JY, Cunningham D, Roth AD, Navarro M, James RD, Karasek P, Jandik P, Iveson T, Carmichael J, Alakl M, Gruia G, Awad L, Rougier P. Irinotecan combined with fluorouracil compared with fluorouracil alone as first-line treatment for metastatic colorectal cancer: a multicentre randomised trial. Lancet. 2000 Mar 25;355(9209):1041-7. doi: 10.1016/s0140-6736(00)02034-1. PMID 10744089
- [Result] Eaden JA, Abrams KR, Mayberry JF. The risk of colorectal cancer in ulcerative colitis: a meta-analysis. Gut. 2001 Apr;48(4):526-35. doi: 10.1136/gut.48.4.526. PMID 11247898
- [Result] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Result] Falcone A, Ricci S, Brunetti I, Pfanner E, Allegrini G, Barbara C, Crino L, Benedetti G, Evangelista W, Fanchini L, Cortesi E, Picone V, Vitello S, Chiara S, Granetto C, Porcile G, Fioretto L, Orlandini C, Andreuccetti M, Masi G; Gruppo Oncologico Nord Ovest. Phase III trial of infusional fluorouracil, leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) compared with infusional fluorouracil, leucovorin, and irinotecan (FOLFIRI) as first-line treatment for metastatic colorectal cancer: the Gruppo Oncologico Nord Ovest. J Clin Oncol. 2007 May 1;25(13):1670-6. doi: 10.1200/JCO.2006.09.0928. PMID 17470860
- [Result] Fearon ER. Molecular genetics of colorectal cancer. Annu Rev Pathol. 2011;6:479-507. doi: 10.1146/annurev-pathol-011110-130235. PMID 21090969
- [Result] Folprecht G, Grothey A, Alberts S, Raab HR, Kohne CH. Neoadjuvant treatment of unresectable colorectal liver metastases: correlation between tumour response and resection rates. Ann Oncol. 2005 Aug;16(8):1311-9. doi: 10.1093/annonc/mdi246. Epub 2005 May 3. PMID 15870084
- [Result] Goldberg RM, Tabah-Fisch I, Bleiberg H, de Gramont A, Tournigand C, Andre T, Rothenberg ML, Green E, Sargent DJ. Pooled analysis of safety and efficacy of oxaliplatin plus fluorouracil/leucovorin administered bimonthly in elderly patients with colorectal cancer. J Clin Oncol. 2006 Sep 1;24(25):4085-91. doi: 10.1200/JCO.2006.06.9039. PMID 16943526
- [Result] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Result] Loupakis F, Cremolini C, Salvatore L, Masi G, Sensi E, Schirripa M, Michelucci A, Pfanner E, Brunetti I, Lupi C, Antoniotti C, Bergamo F, Lonardi S, Zagonel V, Simi P, Fontanini G, Falcone A. FOLFOXIRI plus bevacizumab as first-line treatment in BRAF mutant metastatic colorectal cancer. Eur J Cancer. 2014 Jan;50(1):57-63. doi: 10.1016/j.ejca.2013.08.024. Epub 2013 Oct 15. PMID 24138831
- [Result] Engstrom PF, Arnoletti JP, Benson AB 3rd, Chen YJ, Choti MA, Cooper HS, Covey A, Dilawari RA, Early DS, Enzinger PC, Fakih MG, Fleshman J Jr, Fuchs C, Grem JL, Kiel K, Knol JA, Leong LA, Lin E, Mulcahy MF, Rao S, Ryan DP, Saltz L, Shibata D, Skibber JM, Sofocleous C, Thomas J, Venook AP, Willett C; National Comprehensive Cancer Network. NCCN Clinical Practice Guidelines in Oncology: colon cancer. J Natl Compr Canc Netw. 2009 Sep;7(8):778-831. doi: 10.6004/jnccn.2009.0056. No abstract available. PMID 19755046
- [Result] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720
- See also: CTC V5 — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm
- Available data/document: Informed Consent Form — https://drive.google.com/file/d/1_CG_0wzCH_ZUxWXsfARsyWlcx37fOcRq/view?usp=drive_link